CLINICAL TRIAL: NCT00849186
Title: A Pilot Study of Neoadjuvant SUNITINIB MALATE (Sunitinib) in Patients With Renal Cell Carcinoma Undergoing Nephrectomy
Brief Title: Sunitinib and Surgery in Treating Patients With Localized or Metastatic Kidney Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000634770; P30CA016056 (NIH); RPCI-I-95206
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Results first posted 2015-02-06 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-01

CONDITIONS: Kidney Cancer
Keywords: stage I renal cell cancer; stage II renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Sunitinib; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: sunitinib malate; Procedure: neoadjuvant therapy; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: sunitinib malate — oral
Procedure: neoadjuvant therapy — IV
Procedure: therapeutic conventional surgery — Surgery

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving sunitinib before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This clinical trial is studying the side effects of giving sunitinib before surgery and to see how well it works in treating patients with localized or metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of sunitinib malate in patients with localized or metastatic renal cell carcinoma.
* Determine the safety of surgery after 90 days of treatment with sunitinib malate in these patients.

Secondary

* Determine response of these patients after 90 days of treatment with sunitinib malate.

OUTLINE: Patients receive oral sunitinib malate once daily on days 1-90 in the absence of disease progression or unacceptable toxicity. Patients then undergo radical nephrectomy.

After completion of study treatment, patients are followed for 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed renal cell carcinoma

  * Clinical stage T1b, T2, or T3 tumor with or without nodal or hematogenous metastasis
  * Localized or metastatic disease by renal biopsy
* Primary tumor must be amenable to surgical removal
* No history of or known spinal cord compression or carcinomatous meningitis OR evidence of symptomatic brain or leptomeningeal disease by CT scan or MRI

  * Treated, stable, and asymptomatic brain metastases are allowed

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* ANC ≥ 1,500/mm^3
* Platelets ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN) (≤ 5 times ULN if liver function abnormalities are due to underlying malignancy)
* Total bilirubin ≤ 1.5 times ULN
* Creatinine < 2 mg/dL OR creatinine clearance > 40 mL/min
* Calcium ≤ 10.2 mg/dL
* QTc interval < 500 msec
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 (male)-6 (female) months after completion of study treatment
* No serious intercurrent illness including, but not limited to, any of the following:

  * Clinically significant cardiovascular disease (e.g., uncontrolled hypertension, myocardial infarction, unstable angina)
  * New York Heart Association ≥ class II congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Peripheral vascular disease ≥ grade 2
  * Psychiatric illness/social situations that would limit compliance with study requirements
* None of the following conditions within the past 6 months:

  * Myocardial infarction
  * Severe/unstable angina
  * Coronary/peripheral artery bypass graft
  * Symptomatic congestive heart failure
  * Cerebrovascular accident or transient ischemic attack
  * Pulmonary embolism
* No ongoing cardiac dysrhythmias NCI CTCAE version 3.0 ≥ grade 2
* No hypertension that cannot be controlled by medications (i.e., diastolic blood pressure > 100 mm Hg despite optimal medical therapy)
* No known HIV positivity

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-08; Primary Completion 2009-07 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Willie Underwood, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib Malate (Sunitinib): sunitinib malate: 37.5 mg of daily oral sunitinib is given for 90 days prior to surgery
  neoadjuvant therapy: IV
  therapeutic conventional surgery: Surgery
Period: Overall Study
Arm/Group | Sunitinib Malate (Sunitinib)
Started | 26
Completed | 16
Not Completed | 10
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — not treated | 6
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Sunitinib Malate (Sunitinib)
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.24 (9.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Safety of Sunitinib Malate (SM)
Description: Incident Rate: The proportion of the population who experience a grade 3 or higher endpoint-relevant toxic event within 3 months of the beginning of treatment.
Time Frame: 90 days
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Sunitinib Malate (Sunitinib)
Number analyzed (Participants) | 20
proportion of participants | .350 [.1812 to .5671]

2. Primary Outcome: Safety of Surgery After 90 Days of Treatment With SM
Description: Incident Rate: Intraoperative Complication Rate
Time Frame: 90 days
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Sunitinib Malate (Sunitinib)
Number analyzed (Participants) | 20
proportion of participants | .150 [.0524 to .3604]

3. Secondary Outcome: Response Rate After 90 Days of Treatment With SM
Time Frame: 90 days
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Sunitinib: sunitinib malate: oral
  neoadjuvant therapy: IV
  therapeutic conventional surgery: Surgery
Arm/Group | Sunitinib
Number analyzed (Participants) | 20
proportion of participants | .20 [.0807 to .4160]

ADVERSE EVENTS:
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 7 (7)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8)
White blood cell disorder (Blood and lymphatic system disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 6 (6)
Flatulence (Gastrointestinal disorders) | 4 (4)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8)
Oral discomfort (Gastrointestinal disorders) | 2 (2)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 3 (3)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 12 (13)
Influenza like illness (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Depression postoperative (Injury, poisoning and procedural complications) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 8 (8)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood amylase (Investigations) | 1 (1)
Blood amylase increased (Investigations) | 2 (2)
Blood creatinine (Investigations) | 1 (1)
Blood creatinine decreased (Investigations) | 1 (1)
Lipase (Investigations) | 1 (1)
Lipase increased (Investigations) | 6 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (4)
Hypogeusia (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Arteriovenous fistula operation (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes